CLINICAL TRIAL: NCT06142864
Title: Prevalence of Falls and Associated Factors in Haemodialysis Patients
Acronym: Chute-Hemo
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2023_RIPH_019_Chute-Hemo
Record Dates: First submitted 2023-11-15; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Haemodialysis Patients
Keywords: haemodialysis; falls; haemodialysis patients
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- -"Case" patients: -"Case" patients will be patients reporting at least one fall in the last 6 months.
  Interventions: Other: Data collection
- -"Control" patients: -"Control" patients will be patients reporting no fall in the last 6 months.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data collection

SUMMARY:
In France, falls among the elderly lead to more than 100,000 hospitalisations and more than 10,000 deaths each year. A French study published in October 2020 highlighted 5 profiles of older people who fall. However, this study is only based on falls of people over 65 years of age that required hospitalisation.

In haemodialysis patients, several studies have shown that the incidence of falls ranges from 1.18 to 1.6 falls/patient/year. This population is more likely to be frail, suffer from sarcopenia, have reduced functional capacity and be polymedicated, all of which are associated with an increased risk of falls. Few studies have focused on falls in young patients. In one American study, where the population was predominantly African American (about 62%), 28.4% of patients had at least one fall during follow-up. The number of falls in people aged 45-64 years was similar to that in people aged over 75 years.

In clinical practice, few patients report the occurrence of falls other than those leading to an emergency department visit or hospitalisation, and these falls are even less likely to be recorded in the medical record.

To our knowledge, there are few or no data on falls in haemodialysis patients of all ages in a French population. This lack of knowledge is partly due to an underestimation of the problem associated with under-reporting.

A study of the prevalence of falls in a haemodialysis population of all ages is therefore necessary to determine whether there is an interest in implementing a collective and/or individual prevention programme, possibly depending on the identified risk factors for falls.

DETAILED DESCRIPTION:
The main objective is to describe the prevalence of falls in chronic hemodialysis patients of all ages.

The secondary objective is to study factors associated with the occurrence of falls in chronic hemodialysis patients of all ages

ELIGIBILITY:
Inclusion Criteria:

* aged more than 18
* hemodialysis for more than 3 months,
* Who live at home,
* Who speak and understand French
* Who agree to participate in the study.

Exclusion Criteria:

* aged less than 18
* Living in an institution,
* Who are protected by law (guardianship, curatorship, safeguard of justice),
* Who do not speak and/or understand French
* Who have cognitive problems that prevent them from understanding the specific questions for the study.
* People permanently bedridden

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: haemodialysis patients
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
mechanical fall. | Day 0
  The occurrence of a mechanical fall in the last 6 months (occurrence yes or not) will be sought by specific interrogation of the patient.
  Mechanical falls are defined as falling or slipping on the ground or below the starting position of the subject, involuntarily or awkwardly. Falls related to a violent flare-up, loss of consciousness, sudden onset of paralysis as in a stroke or seizure of epilepsy are not considered.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Ufr Medecine Urca, Reims
  - Université de Reims Champagne Ardenne, Reims

IPD SHARING:
Plan to Share IPD: Undecided